CLINICAL TRIAL: NCT01707771
Title: Effect of Gastric Bypass Versus Diet on Cardiovascular Risk Factors
Brief Title: Bariatric Surgery and HDL-cholesterol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Geltrude Mingrone, Professor, Catholic University of the Sacred Heart
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HDL-2008
Record Dates: First submitted 2012-10-10; First posted 2012-10-16 (Estimated); Last update posted 2012-10-16 (Estimated); Status verified 2012-10

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid | interventions — Gastric Bypass; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Roux-en-Y gastric bypass (Active Comparator): Both sexes, age between 30 and 60 years, BMI =/> 35 kg/m2
  Interventions: Procedure: Roux-en-Y gastric bypass
- diet and lifestyle modifications (Active Comparator): Both sexes, age between 30 and 60 years, BMI =/> 35 kg/m2
  Interventions: Behavioral: diet and lifestyle modifications

INTERVENTIONS:
Procedure: Roux-en-Y gastric bypass — Active Comparator: Roux-en-Y gastric bypass
  Arms: Roux-en-Y gastric bypass
Behavioral: diet and lifestyle modifications — Active Comparator: diet and lifestyle modifications
  Arms: diet and lifestyle modifications

SUMMARY:
Objective: to assess the effect of gastric bypass on HDL-cholesterol concentration and its Apolipoprotein A4 content at 1 year following bariatric surgery in comparison with a hypocaloric diet. Secondary aim was to measure total cholesterol and triglycerides levels as well as insulin sensitivity after interventions.

Summary Background Data: Very few prospective uncontrolled studies have investigated the effects of Roux-en-Y gastric bypass (RYGB) on cardiovascular risk factors. No controlled studies had as primary goal the changes in HDL-cholesterol after gastric bypass.

Methods: Forty subjects with a BMI>40 or ≥35 kg/m2 in the presence of diabetes were enrolled.

Twenty of them were operated of RYGB while 20 received lifestyle modification suggestions and medical therapy for obesity complications (diabetes, hypertension and hyperlipidemia).

DETAILED DESCRIPTION:
Study design The study was an unblinded, prospective, non randomized clinical trial. Participants were recruited from referrals for treatment of morbid obesity between September 2008 and July 2009. One year follow-up was completed in September 2011.

The aim of the study related to the changes in HDL-cholesterol at 1 year after the intervention. Secondary aims were the changes in Apolipoprotein 4 (Apo4) and insulin sensitivity after the interventions.

Twenty morbidly-obese subjects (11 women and 9 men), whose 14 with normal glucose tolerance and 6 with type 2 diabetes mellitus (T2DM), have been studied before and 1, 2, 3, 6, 9 and 12 months after bariatric surgery.

Twenty morbidly-obese subjects (12 women and 8 men), 15 with normal glucose tolerance and 5 with T2DM, in the waiting list for bariatric surgery were enrolled in the protocol and underwent medical therapy for obesity complications (diabetes, hypertension and hyperlipidemia) and lifestyle modification suggestions.

Participants were eligible for inclusion if they had a BMI of 40 kg/m2 or >35 kg/m2 in presence of type 2 diabetes, were aged 30 to 60 years, and had not sustained weight loss in the previous 1 year. Exclusion criteria were a history of major abdominal or bariatric surgery, disabling cardiac or pulmonary diseases, cancer, long-term treatment with oral corticosteroids, and mental illness.

Roux-&-Y Gastric Bypass (RYGB) involves the use of a surgical stapler to create a small and vertically oriented gastric pouch with a volume usually < 30 ml. The upper pouch is completely divided by the gastric remnant and is anastomosed to the jejunum, 75 cm distally to the Treitz's ligament , through a narrow gastrojejunal anastomosis in a Roux-en-Y fashion. Bowel continuity is restored by an entero-entero anastomosis, between the excluded biliary limb and the alimentary limb, performed at 150 cm from the gastrojejunostomy.

Lifestyle modifications A hypocaloric diet (15 kcal/kgbw containing 55% carbohydrates, 30% lipids and 15% proteins) was prescribed together with the indications to perform 30 minutes brisk walk each day. Patients had open access to a diabetologist every 3 months. Medical therapies, including pharmaceutical agents, were assigned on an individual basis.

Anthropometric measures Body weight was measured to the nearest 0.1 kg with a beam scale and height to the nearest 0.5 cm using a stadiometer (Holatin, Crosswell, Wales, U.K.).

Blood pressure Blood pressure was measured 3 times with an appropriately sized cuff after the participant had rested for 5 minutes, and the last 2 measurements were averaged.

Oral glucose tolerance test A standard 75-g oral glucose tolerance test (OGTT) was performed after an overnight fasting with blood sampling at 0, 30, 60, 90, 120, and 180 min. Samples were placed in chilled tubes, and plasma was separated within 20 min and stored at -80°C.

Analytical methods Blood was drawn in the morning after an overnight fast. The sera and plasma were immediately separated by centrifugation at 4°C and stored at -80°C until assay.

Plasma glucose was measured by the glucose-oxidase method (Beckman, Fullerton, CA). Plasma insulin was assayed by microparticle-enzyme immunoassay (Abbott, Pasadena, CA) with a sensitivity of 1 μU/ml and an intra-assay CV of 6.6%.

Total cholesterol and triglycerides were measured enzymatically. HDL-cholesterol was measured after precipitating apolipoprotein B-containing lipoproteins with dextran sulfate and magnesium chloride.

HbA1c serum levels were measured by high-performance liquid-chromatography (normal range 3.5-6.5%) Apo A4 was assessed by ELISA (Cusabio Biotech, Wuhan, Hubei, China); the detection range is from 15.62 μg/l to 1000 μg/l and the minimum detectable concentration is 4 μg/l.

Insulin Sensitivity Models

The OGTT and fasting plasma glucose and insulin were used to compute the insulin sensitivity. Insulin resistance was assessed using the homeostasis model assessment (HOMA-IR) originally described by Mathew et al. HOMA-IR was calculated using the following equation:

HOMA-IR(μU/ml∙mg/dl)=fasting insulin(μU/ml)∙(fasting glucose (mg/dl))/405 Peripheral insulin sensitivity was assessed by the Oral Glucose Insulin Sensitivity (OGIS) model. OGIS is an index of insulin sensitivity calculated in this case from the 3 hours OGTT and it is an estimate of the glucose clearance during a hyperinsulinemic euglycemic glucose clamp expressed in ml/min per square meter of body surface area.

Statistics All of the data are expressed as means ± SD unless otherwise specified. The Wilcoxon paired-sample test was used for intragroup comparisons. Two-sided P < 0.05 was considered significant. Nonparametric Spearman correlations were used to assess linear relationships between single variables.

We calculated that a total of 30 participants would give 80% power to detect a significant (P < 0.05) difference between the groups. To allow for possible dropouts and add power for analysis of secondary outcomes, we decided to enroll 40 participants.

ELIGIBILITY:
Inclusion Criteria:

* BMI =/> 35 kg/m2,
* age 30-60 years,
* both sexes

Exclusion Criteria:

* history of major abdominal or bariatric surgery,
* disabling cardiac or pulmonary diseases,
* cancer,
* long-term treatment with oral corticosteroids, and
* mental illness

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2008-09; Primary Completion 2011-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
changes in HDL-cholesterol Baseline to 1 year HDL-cholesterol changes: baseline to 1 year | 1 year

SECONDARY OUTCOMES:
changes in Apolipoprotein 4 (Apo4) and insulin sensitivity | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Geltrude Mingrone, MD, Principal Investigator — Catholic University
Locations (1):
- Catholic University, Rome, Italy

REFERENCES:
- [Derived] Raffaelli M, Guidone C, Callari C, Iaconelli A, Bellantone R, Mingrone G. Effect of gastric bypass versus diet on cardiovascular risk factors. Ann Surg. 2014 Apr;259(4):694-9. doi: 10.1097/SLA.0b013e31829d6989. PMID 23979288